CLINICAL TRIAL: NCT06331650
Title: A Single-arm Pilot Study of First-line Treatment With Carbognilumab Combined With Chemotherapy in Patients With STK11-mutated Advanced or Postoperative Recurrent Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC202314
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadonilimab (Experimental)
  Interventions: Drug: cadonilimab

INTERVENTIONS:
Drug: cadonilimab — Cardunnilizumab: the recommended dose is 10mg/kg every 3 weeks on the first day of each cycle; Discontinuation of the drug may be considered if intolerable adverse reactions occur.

SUMMARY:
To evaluate the safety and tolerability of carbognilumab combined with chemotherapy as the first-line treatment for patients with STK11 mutated advanced or postoperative recurrent non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. voluntary participation in clinical research; Fully understand and Informed the study and sign the Informed Consent Form (ICF); Be willing to follow and be able to complete all trial procedures.
2. Age ≥18 years old and ≤75 years old when signing ICF.
3. histologically or cytologically confirmed advanced or postoperative recurrent non-small cell lung cancer (AJCC 8th edition).
4. STK11 mutations were detected by NGS, and no other sensitive mutations could be targeted therapy (including EGFR, ALK, ROS1, RET, c-Met, HER2, BRAF gene rearrangement, fusion, amplification, and skipping).
5. The patient had not received systemic antitumor therapy.
6. Patients who had received one prior chemotherapy regimen were allowed, regardless of whether chemotherapy was administered before, after, or concurrently with targeted therapy.
7. Patients receiving adjuvant or neoadjuvant therapy were allowed if adjuvant/neoadjuvant therapy had been completed at least 12 months before diagnosis of advanced or postoperative recurrent NSCLC.
8. The interval between the end of previous nonsystemic antitumor therapy and the start of study medication had to be 4 weeks or more. Treatment-related AE recovered to CTCAE 4.03≤ grade 1 (except grade 2 alopecia).
9. have at least one measurable target lesion as assessed by the investigator according to iRECIST requirements within 4 weeks before enrollment.
10. If available, patients can provide eligible tumor tissue for PD-L1 expression level measurement.
11. an ECOG PS score of 0 or 1 within 7 days before the first dose of study medication.
12. predicted survival time ≥12 weeks (3 months).
13. had good major organ function, defined as meeting the following criteria, and had not received blood transfusions, albumin, recombinant human thrombopoietin, or colony-stimulating factor (CSF) within 14 days before the first dose of study medication.
14. Female patients must meet one of the following conditions:

1) menopause, defined as absence of menses for at least 1 year and no confirmed cause other than menopause, or (2) having undergone sterilization (removal of ovaries and/or uterus) 3) be fertile, provided that: Patients had to have a negative serum pregnancy test within 7 days before randomization and agree to use contraception with an annual failure rate of <1% or to abstain from heterosexual intercourse for at least 120 days from the date of written informed consent until the last dose of trial drug was administered. At least 150 days after the last dose of chemotherapy) (contraceptive methods with an annual failure rate of <1% include bilateral tubal ligation, male sterilization, proper use of ovulation-suppressing hormonal contraceptives, hormone-releasing intrauterine devices, and copper intrauterine devices or condoms), and Do not breastfeed.

15.Male patients had to agree to either abstain from sex (avoid heterosexual intercourse) or to use contraception, as specified by either abstinence or use of condoms to prevent exposure of the drug to the embryo during chemotherapy (paclitaxel/pemetrexed/carboplatin) for the duration of treatment with a woman of reproductive age or a pregnant partner and for at least 150 days after the last dose of chemotherapy. Regular abstinence (e.g., calendar day, ovulation, basal body temperature, or postovulatory methods of contraception) and in vitro ejaculation are ineligible methods of contraception.

Exclusion Criteria:

1. received systemic therapy for advanced NSCLC within 4 weeks after enrollment;
2. the subjects had a history or concurrent history of other malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix).
3. candidates for or prior recipients of organ or bone marrow transplantation.
4. uncontrollable pleural, pericardial, or ascites with appropriate interventions.
5. subjects with clinically symptomatic CNS metastases (e.g., brain edema, need for hormonal intervention, or progression of brain metastases). Patients who had received previous treatment for brain or meningeal metastases were eligible if they had been clinically stable (on MRI) for at least 2 months and had stopped systemic hormone therapy (at a dose of >10mg per day of prednisone or other iso-efficacy hormones) for more than 2 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety assessments and ORR | 2 years
  Objective response rate (ORR) as assessed by investigators according to iRECIST in patients with STK11-mutated advanced or postoperative recurrent non-small cell lung cancer treated with carbognilumab plus chemotherapy as first-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: zhou chengzhi, doctor, Principal Investigator — Principal Investigator
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangdong, Guangzhou, China